CLINICAL TRIAL: NCT02353520
Title: "Reliability of Motricity Index Strength Assessments for Upper Extremity in Post Stroke Hemiparesis- a Correlation Study''
Status: Completed | Type: Observational
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, ASHIMA ARORA, ASHIMA ARORA, Maharishi Markendeswar University (Deemed to be University)
Other Study IDs: RELIBILITY OF MOTRICITY INDEX
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: motricity index strength assessment

SUMMARY:
Initially, a written consent was obtained from each participant. Then they became familiar with the procedure. For intrarater reliability, the first rater assessed the strength of pinch grip, elbow flexion and shoulder abduction in three different sessions at short intervals on same day in same environmental conditions. All the assessments were performed on the same day in three sessions. Assessment duration of all the sessions was 5 minutes.

For inter-rater reliability, Before the beginning of Procedure both the raters were familiarized with the motricity index. The motricity index was administered by two different raters on the same subjects within 2 days who were blind to each others results and heir results were recorded separately.

DETAILED DESCRIPTION:
Initially, a written consent was obtained from each participant. Then they became familiar with the procedure. For intrarater reliability, the first rater assessed the strength of pinch grip, elbow flexion and shoulder abduction in three different sessions at short intervals on same day in same environmental conditions. All the assessments were performed on the same day in three sessions. Assessment duration of all the sessions was 5 minutes.

For inter-rater reliability, Before the beginning of Procedure both the raters were familiarized with the motricity index. The motricity index was administered by two different raters on the same subjects within 2 days who were blind to each others results and heir results were recorded separately.

PATIENT POSITION The patient was sitting on a chair or on the edge of the bed, but can be tested lying supine if necessary. In the arm the three movements tested were pinch grip, elbow flexion and shoulder abduction.

Pinch grip Assessed by asking the patient to grip a 2.5 cm cube between the thumb and fore finger. The object was on a flat surface (for example, a book).

The tester scored contraction of any forearm or small hand muscles as follows:

0 No movement. 11 Beginnings of prehension (any movement of finger or thumb). 19 Able to grip the cube, but not hold it against gravity (examiner may need to lift the wrist) 22 Able to grip and hold the cube against gravity, but not against a weak pull.

26 Able to grip and hold the cube against a weak pull, but weaker than the other side.

33 Normal pinch grips. Elbow flexion The elbow was tested with the elbow flexed to 90°, forearm horizontal and upper arm vertical. The patient was asked to bend the elbow so that the hand touches the shoulder. The examiner resisted with a hand on the wrist, and monitored the biceps. If there was no movement, the examiner holded the elbow out so that the arm was horizontal, and gave a score of 14 if movement was then seen.

Shoulder abduction The elbow was fully flexed and against the chest and the patient was asked to abduct the arm. The examiner monitored contraction of the deltoid movement of shoulder girdle does not count-there must be movement of humerus in relation to scapula). A score of 19 was given when the shoulder was abducted to more than 90◦ beyond the horizontal against gravity but not against resistance.

According to the quality of muscle contraction the score was recorded. Rater was also aware of any trick motion such as leaning the back during the movement by placing one hand on their back. Finally, all three scores were summed and the Motricity Index for upper extremity was calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Post stroke hemiparetic patients were included in the study.
2. Age 37 to 76 years.
3. Mini mental status examination score ≥ 23.
4. Individuals having Brunnstrom stage 4 and 5 in upper extremity.
5. Individuals should not be taking any physiotherapy treatment for stroke

Exclusion Criteria:

1. Patients at the acute or chronic commonly seen at clinics.
2. Patient having any musculo-skeletal disorder in upper limb.
3. Patient having any trauma on their upper extremity.
4. Patient having any neurological disorder other than stroke.
5. Any hypersensitivity or hyposensitivity disorder

Ages: 37 Years to 76 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients of both sex
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Motricity index strength assessment | 1 month
  Initially, a written consent was obtained from each participant. Then they became familiar with the procedure. For intrarater reliability, the first rater assessed the strength of pinch grip, elbow flexion and shoulder abduction in three different sessions at short intervals on same day in same environmental conditions. All the assessments were performed on the same day in three sessions. Assessment duration of all the sessions was 5 minutes.
  For inter-rater reliability, Before the beginning of Procedure both the raters were familiarized with the motricity index. The motricity index was administered by two different raters on the same subjects within 2 days who were blind to each others results and heir results were recorded separately.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Senthil P Kumar, PhD, Study Director — MMIPR